CLINICAL TRIAL: NCT06114628
Title: A Seamless Phase 2B/C Platform Trial to Evaluate Multiple Regimens and Durations of Treatment in Pulmonary Tuberculosis
Brief Title: Platform Assessing Regimens and Durations In a Global Multisite Consortium for TB
Acronym: PARADIGM4TB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Radboud University Medical Center (Other); London School of Hygiene and Tropical Medicine (Other); University of Oxford (Other); Research Center Borstel (Other); Lygature (Unknown); TASK Applied Science (Other); Vita-Salute San Raffaele University (Unknown); Helmholtz Zentrum Munchen (Unknown); KNCV Tuberculosis Foundation (Other); Critical Path Institute (Unknown); European Lung Foundation (Unknown); Instituto de Saude Publica da Universidade do Porto (Other); University of Liverpool (Other); Institut de Recherche pour le Developpement (Other Government); University of Hamburg-Eppendorf (Other); University of California, San Francisco (Other); TB Alliance (Unknown); Find (Other); University of Milano (Unknown); University of St Andrews (Other); Uppsala University (Other); European Respiratory Society (Other); Tuberculosis Network European Trialsgroup (Network); Janssen, LP (Industry); Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry); German Center for Infection Research (Other); LMU University Hospital Munich (Unknown); University of Cambridge (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNITE4TB-01
Record Dates: First submitted 2023-10-17; First posted 2023-11-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — GSK656; 2-(2-methyl-1,4-dioxa-8-azaspiro(4.5)dec-8-yl)-8-nitro-6-(trifluoromethyl)-4H-1,3-benzothiazin-4-one; bedaquiline; OPC-67683; Fumigant 93; pretomanid; Moxifloxacin; Linezolid; Pyrazinamide; Rifampin; Isoniazid; Protons; Ethambutol; delpazolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- A. Standard TB Regimen. 2HRZE/4HR (Active Comparator): 24 weeks treatment in both Phase 2B and 2C - 8 weeks Rifampicin, Isoniazid, Pyrazinamide, Ethambutol followed by 16 weeks Rifampicin and Isoniazid.
  Interventions: Drug: Pyrazinamide (Z); Drug: Rifampicin (R); Drug: Isoniazid (H); Drug: Ethambutol (E)
- Arm B. BDM (Experimental): Bedaquiline, Delamanid, Moxifloxacin for 16 weeks in Phase 2B
  Interventions: Drug: Bedaquiline (B); Drug: Delamanid (D); Drug: Moxifloxacin (M)
- Arm C. BDM + Gan (Experimental): Bedaquiline, Delamanid, Moxifloxacin and Ganfeborole for 16 weeks in Phase 2B Bedaquiline, Delamanid, Moxifloxacin and Ganfeborole for 8-16 weeks in phase 2C
  Interventions: Drug: Ganfeborole; Drug: Bedaquiline (B); Drug: Delamanid (D); Drug: Moxifloxacin (M)
- Arm D. BDZ + Gan (Experimental): Bedaquiline, Delamanid, Pyrazinamide and Ganfeborole for 16 weeks in Phase 2B Bedaquiline, Delamanid, Pyrazinamide and Ganfeborole for 8-16 weeks in phase 2C
  Interventions: Drug: Ganfeborole; Drug: Bedaquiline (B); Drug: Delamanid (D); Drug: Pyrazinamide (Z)
- Arm E. BDL + 656 (Experimental): Bedaquiline, Delamanid, Linezolid and Ganfeborole for 8 weeks followed by 8 weeks Bedaquiline, Delamanid and Ganfeborole in Phase 2B Bedaquiline, Delamanid, Linezolid and Ganfeborole for 8 weeks followed by 0-8 weeks Bedaquiline, Delamanid and Ganfeborole in Phase 2C
  Interventions: Drug: Ganfeborole; Drug: Bedaquiline (B); Drug: Delamanid (D); Drug: Linezolid (L)
- Arm F. BPaM + Gan (Experimental): Bedaquiline, Pretomanid, Moxifloxacin and Ganfeborole for 16 weeks in Phase 2B Bedaquiline, Pretomanid, Moxifloxacin and Ganfeborolefor 8-16 weeks in Phase 2C
  Interventions: Drug: Ganfeborole; Drug: Bedaquiline (B); Drug: Pretomanid (Pa); Drug: Moxifloxacin (M)
- Arm G. BDM + BTZ-043 (Experimental): Bedaquiline, Delamanid, Moxifloxacin and BTZ-043 for 16 weeks in Phase 2B Bedaquiline, Delamanid, Moxifloxacin and BTZ-043 for 8-16 weeks in phase 2C
  Interventions: Drug: BTZ-043; Drug: Bedaquiline (B); Drug: Delamanid (D); Drug: Moxifloxacin (M)
- Arm H. BDZ + BTZ-043 (Experimental): Bedaquiline, Delamanid, Pyrazinamide and BTZ-043 for 16 weeks in Phase 2B Bedaquiline, Delamanid, Pyrazinamide and BTZ-043 for 8-16 weeks in phase 2C
  Interventions: Drug: BTZ-043; Drug: Bedaquiline (B); Drug: Delamanid (D); Drug: Pyrazinamide (Z)
- Arm I. BDL + BTZ-043 (Experimental): Bedaquiline, Delamanid, Linezolid and BTZ-043 for 8 weeks followed by 8 weeks Bedaquiline, Delamanid and BTZ-043 in Phase 2B Bedaquiline, Delamanid, Linezolid and BTZ-043 for 8 weeks followed by 0-8 weeks Bedaquiline, Delamanid and BTZ-043 in Phase 2C
  Interventions: Drug: BTZ-043; Drug: Bedaquiline (B); Drug: Delamanid (D); Drug: Linezolid (L)
- Arm J. BPaM + BTZ-043 (Experimental): Bedaquiline, Pretomanid, Moxifloxacin and BTZ-043 for 16 weeks in Phase 2B Bedaquiline, Pretomanid, Moxifloxacin and BTZ-043 for 8-16 weeks in Phase 2C
  Interventions: Drug: BTZ-043; Drug: Bedaquiline (B); Drug: Pretomanid (Pa); Drug: Moxifloxacin (M)
- Arm K. BMZ + BTZ-043 (Experimental): Bedaquiline, Moxifloxacin, Pyrazinamide and BTZ-043 for 16 weeks in Phase 2B Bedaquiline, Moxifloxacin, Pyrazinamide and BTZ-043 for 8-16 weeks in phase 2C
  Interventions: Drug: BTZ-043; Drug: Bedaquiline (B); Drug: Moxifloxacin (M); Drug: Pyrazinamide (Z)
- Arm L. BD + Gan + BTZ-043 (Experimental): Bedaquiline, Delamanid, Ganfeborole and BTZ-043 for 16 weeks in Phase 2B Bedaquiline, Delamanid, Ganfeborole and BTZ-043 for 8-16 weeks in phase 2C
  Interventions: Drug: Ganfeborole; Drug: BTZ-043; Drug: Bedaquiline (B); Drug: Delamanid (D)
- Arm M: BDM + Q (Experimental): Bedaquiline, delamanid, moxifloxacin, quabodepistat for 16 weeks in Phase 2B
  Interventions: Drug: Bedaquiline (B); Drug: Delamanid (D); Drug: Moxifloxacin (M); Drug: Quabodepistat (Q)
- Arm N: BPAM + Q (Experimental): Bedaquiline, pretomanid, moxifloxacin, quabodepistat for 16 weeks in Phase 2B
  Interventions: Drug: Bedaquiline (B); Drug: Pretomanid (Pa); Drug: Moxifloxacin (M); Drug: Quabodepistat (Q)
- Arm O: BD + Gan + Q (Experimental): Bedaquiline, delamanid, ganfeborole, quabodepistat for 16 weeks in Phase 2B
  Interventions: Drug: Ganfeborole; Drug: Bedaquiline (B); Drug: Delamanid (D); Drug: Quabodepistat (Q)
- Arm P: BPa + Gan +Q (Experimental): Bedaquiline, pretomanid, ganfeborole, quabodepistat for 16 weeks in Phase 2B
  Interventions: Drug: Ganfeborole; Drug: Bedaquiline (B); Drug: Pretomanid (Pa); Drug: Quabodepistat (Q)
- Arm Q: BPa + DZD + BTZ-043 (Experimental): Bedaquiline, pretomanid, delpazolid, BTZ-043 for 16 weeks in Phase 2B
  Interventions: Drug: BTZ-043; Drug: Bedaquiline (B); Drug: Pretomanid (Pa); Drug: Delpazolid (DZD)

INTERVENTIONS:
Drug: Ganfeborole — Oral daily dosage of 20mg.
  Other Names: GSK3036656
  Arms: Arm C. BDM + Gan; Arm D. BDZ + Gan; Arm E. BDL + 656; Arm F. BPaM + Gan; Arm L. BD + Gan + BTZ-043; Arm O: BD + Gan + Q; Arm P: BPa + Gan +Q
Drug: BTZ-043 — Oral daily dosage of 1000mg.
  Arms: Arm G. BDM + BTZ-043; Arm H. BDZ + BTZ-043; Arm I. BDL + BTZ-043; Arm J. BPaM + BTZ-043; Arm K. BMZ + BTZ-043; Arm L. BD + Gan + BTZ-043; Arm Q: BPa + DZD + BTZ-043
Drug: Bedaquiline (B) — Oral daily dosage of 400mg for the first 2 weeks, thereafter 100mg daily until end of treatment.
  Arms: Arm B. BDM; Arm C. BDM + Gan; Arm D. BDZ + Gan; Arm E. BDL + 656; Arm F. BPaM + Gan; Arm G. BDM + BTZ-043; Arm H. BDZ + BTZ-043; Arm I. BDL + BTZ-043; Arm J. BPaM + BTZ-043; Arm K. BMZ + BTZ-043; Arm L. BD + Gan + BTZ-043; Arm M: BDM + Q; Arm N: BPAM + Q; Arm O: BD + Gan + Q; Arm P: BPa + Gan +Q; Arm Q: BPa + DZD + BTZ-043
Drug: Delamanid (D) — Oral daily dosage of 300mg.
  Arms: Arm B. BDM; Arm C. BDM + Gan; Arm D. BDZ + Gan; Arm E. BDL + 656; Arm G. BDM + BTZ-043; Arm H. BDZ + BTZ-043; Arm I. BDL + BTZ-043; Arm L. BD + Gan + BTZ-043; Arm M: BDM + Q; Arm O: BD + Gan + Q
Drug: Pretomanid (Pa) — Oral daily dosage of 200mg.
  Arms: Arm F. BPaM + Gan; Arm J. BPaM + BTZ-043; Arm N: BPAM + Q; Arm P: BPa + Gan +Q; Arm Q: BPa + DZD + BTZ-043
Drug: Moxifloxacin (M) — Oral daily dosage of 400mg.
  Arms: Arm B. BDM; Arm C. BDM + Gan; Arm F. BPaM + Gan; Arm G. BDM + BTZ-043; Arm J. BPaM + BTZ-043; Arm K. BMZ + BTZ-043; Arm M: BDM + Q; Arm N: BPAM + Q
Drug: Linezolid (L) — Oral daily dosage of 600mg for the first 8 weeks.
  Arms: Arm E. BDL + 656; Arm I. BDL + BTZ-043
Drug: Pyrazinamide (Z) — Oral daily dosage of 1200mg-2000mg depending on weight.
  Arms: A. Standard TB Regimen. 2HRZE/4HR; Arm D. BDZ + Gan; Arm H. BDZ + BTZ-043; Arm K. BMZ + BTZ-043
Drug: Rifampicin (R) — Oral daily dosage of 450mg-750mg depending on weight.
  Arms: A. Standard TB Regimen. 2HRZE/4HR
Drug: Isoniazid (H) — Oral daily dosage of 225mg-375mg depending on weight.
  Arms: A. Standard TB Regimen. 2HRZE/4HR
Drug: Ethambutol (E) — Oral daily dosage of 825mg-1375mg depending on weight.
  Arms: A. Standard TB Regimen. 2HRZE/4HR
Drug: Delpazolid (DZD) — Oral daily dosage of 1200mg
  Arms: Arm Q: BPa + DZD + BTZ-043
Drug: Quabodepistat (Q) — Oral daily dosage of 30mg
  Arms: Arm M: BDM + Q; Arm N: BPAM + Q; Arm O: BD + Gan + Q; Arm P: BPa + Gan +Q

SUMMARY:
The UNITE4TB consortium is a group of universities and pharmaceutical companies funded by the European Union. This consortium are carrying out a trial to find better and faster ways to treat tuberculosis (TB). The standard treatment for TB takes 24 weeks and uses four drugs. The consortium want to find new treatments that are faster but just as safe and effective.

In the trial, two new drugs will be used, BTZ-043 and GSK3036656, along with the drugs that are already used to treat TB in a variety of combinations (11 different combinations initially). These new drugs have worked well in tests with animals and have reduced the amount of TB bacteria in people's sputum/phlegm when used alone for two weeks. These new drugs will be used in combination with other TB drugs for a longer time (up to 16 weeks) in people with TB. The UNITE4TB consortium want to see if they work well and are safe.

This trial will take place at sites across the world and will involve people with TB of the lungs that would usually respond well to the standard treatment. But the new treatments being tested might also work for people with drug resistant TB, that's harder to treat.

The trial has two parts. In the first part, different combinations of drugs will be tried on up to 700 people for 16 weeks. These combinations will be compared to the standard 24-week treatment to see which ones work the best and are safe.

In the second part, the best combinations from the first part will be taken to try to find out what the best length of time is to give the treatment for. These combinations will be tried on up to 1800 people giving them either 8, 10, 12, 14 or 16 weeks treatment. The investigators will follow these people for a total of 72 weeks to make sure the treatment is working.

The UNITE4TB consortium hope that this trial will find new treatments that are fast, safe, and effective for both regular TB and resistant TB. If it works, it can then be tested again in a bigger trial to be sure.

DETAILED DESCRIPTION:
Study Design:

This will be a randomised, open-label, multicentre, seamless phase 2B (regimen selection) and 2C (duration randomisation), multi-arm multi-stage, platform clinical trial

Overall objective:

The overall objective is to identify novel drug regimen(s) with acceptable safety profile, non-inferior efficacy, and shortened treatment duration compared to the standard-of-care 24-week HRZE/HR regimen (isoniazid + rifampicin + pyrazinamide + ethambutol for 8 weeks then isoniazid + rifampicin for 16 weeks) that could be used to treat both rifampicin-susceptible and resistant TB.

Specific sub-objectives:

The objective of the Phase 2B stage is to identify novel regimens of 16 weeks' duration with acceptable safety profile and the greatest potential, based on assessment of quantitative sputum liquid culture and treatment failure/relapse, to progress to investigation of optimal treatment duration

Amongst the regimens selected for progression from phase 2B to phase 2C stage, the objective is then to further evaluate the safety profile of these regimens and to identify the optimal treatment duration (between 8 and 16 weeks) based on unfavourable outcome to support advancement to future Phase 3 trials.

Setting:

Specialist TB clinics and research centres in sites across Europe, Asia, Africa and South America

Population:

Adults with newly diagnosed, rifampicin-susceptible pulmonary TB

Duration:

Individual participant participation will be for 72 weeks. The total duration of trial is 5 years.

Interventions:

Phase 2B: Participants will be randomised (1:1:1..1) to the following 12 arms (A-L) initially. Additional arms maybe added through protocol amendment.

Control, standard-of-care regimen, given for 24 weeks

A. Isoniazid + rifampicin + pyrazinamide + ethambutol for 8 weeks then isoniazid + rifampicin for 16 weeks

Novel treatment regimens each given for 16 weeks

B. Bedaquiline + delamanid + moxifloxacin

C. Bedaquiline + delamanid + moxifloxacin + GSK306656

D. Bedaquiline + delamanid + pyrazinamide + GSK306656

E. Bedaquiline + delamanid + linezolid (for first 8 weeks) + GSK306656

F. Bedaquiline + pretomanid + moxifloxacin + GSK306656

G. Bedaquiline + delamanid + moxifloxacin + BTZ-043

H. Bedaquiline + delamanid + pyrazinamide + BTZ-043

I. Bedaquiline + delamanid + linezolid (for first 8 weeks) + BTZ-043

J. Bedaquiline + pretomanid + moxifloxacin + BTZ-043

K. Bedaquiline + moxifloxacin + pyrazinamide + BTZ-043

L. Bedaquiline + delamanid + GSK306656 + BTZ-043

There are two planned interim analyses of safety and efficacy data by an Independent Data Monitoring Committee in Phase 2B. The first interim analysis will occur when the last participant for arms to be included in the analysis, completes 16 weeks of treatment and all necessary data are available. The second interim analysis will occur when the last participant for arms to be included in the analysis completes to week 48 (from randomisation) and all necessary data are available. The IDMC will make recommendation to the Trial Steering Committee (TSC) and Asset Holders on the progression of regimens to Phase 2C. The TSC will make the final decision. Arm B (bedaquiline + delamanid + moxifloxacin) will not be considered for progression to 2C.

Phase 2C:

For regimens selected for progression (following interim phase 2B evaluation). Participants will be randomised to treatment durations of either 8 weeks, 10 weeks, 12 weeks, 14 weeks, 16 weeks or to the 24-week standard-of-care regimen (as described above).

Primary Efficacy Outcome Measure(s) -

Phase 2B: rate of change in log10(TTP) over 0 to 12 weeks, where TTP is time to positivity measured in days from MGIT culture

Phase 2C: Favourable/unfavourable status (binary) at week 48 from randomisation

Safety Outcome Measures (Phase 2B and 2C) -

The following outcomes will be reported up to week 26 from randomisation (unless otherwise stated):

* Grade 3/4/5 adverse events (DAIDS grading scale)
* Serious Adverse Events
* Adverse Events of Special Interest
* Regimen-related adverse events leading to withdrawal from the study
* Adverse events leading to discontinuation of the regimen

Number of Participants to be Studied:

Up to 2500 overall - 700 in phase 2B and 1800 in phase 2C (distribution between phases depends on progression according to specified decision-making steps)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above at screening (or above age of legal consent at screening, if this is higher than 18 years in the jurisdiction in which the study is taking place)
2. Clinical evidence of active TB disease, meeting either or both of the following criteria:

   * Symptoms consistent with pulmonary TB at screening AND/OR
   * Imaging findings consistent with active pulmonary TB on chest X-ray performed at screening or within 7 days prior to screening
3. At least one sputum specimen produced at screening tested on Xpert MTB/RIF Ultra that has:

   * a semi-quantitative result of 'medium' or 'high' AND
   * does not show rifampicin resistance
4. Body weight within the range of 30 to 100kg and body mass index within the range of 15 to 40kg/m2
5. Willing to comply with study visits, all study procedures and treatment observation
6. Resident at a fixed address that is readily accessible for visiting, within feasible travelling distance to the site and likely to remain resident there for the duration of trial follow-up
7. Has provided written informed consent

Exclusion Criteria:

1. Taken more than 1 daily dose of medication with anti-tuberculous activity during the 14 days prior to randomisation (isoniazid, rifampicin, pyrazinamide, ethambutol; linezolid, moxifloxacin, levofloxacin or amikacin) (for Phase 2b and Phase 2c)
2. Known isoniazid resistance (at sites where national isoniazid monoresistance is greater than 10% rapid testing at screening is mandated; at other sites rapid testing at screening is optional)
3. Known or suspected extra-thoracic TB, miliary TB or disseminated TB (in the judgement of the investigator; note uncomplicated pleural effusion occupying <50% of hemithorax or concomitant intra- or extra-thoracic lymphadenopathy are not exclusions)
4. Severe clinical pulmonary TB e.g. respiratory failure or complications likely to require hospital admission in the opinion of the investigator
5. Poor general condition (Karnofsky score ≤50) OR where any delay in treatment cannot be tolerated in the opinion of the investigator
6. Active malignancy requiring systemic therapy, radiotherapy or palliative therapy
7. History of myocardial infarction, coronary heart disease or congestive cardiac failure; long QT syndrome or clinically significant arrhythmias; pulmonary hypertension; any known congenital cardiac problems; family history of long QT syndrome or sudden death from unknown or cardiac related cause; uncontrolled arterial hypertension (not excluded if this is corrected prior to randomisation)
8. Vitiligo
9. History of seizure(s)
10. Current tendinitis (any cause) or history of tendinopathy associated with fluoroquinolone use
11. History of vascular aneurysm
12. Symptomatic peripheral neuropathy causing greater than minimal interference with usual social and functional activities
13. Current alcohol or illicit drug use sufficient to compromise the safety of the participant or research staff or compromise adherence to study procedures, in the opinion of the investigator
14. Any current or recent use of amphetamines or methamphetamines, either reported or evident on toxicity screen, if performed
15. Any other medically or socially significant condition (e.g. psychiatric illness, chronic diarrhoeal disease, metabolic condition, other cardiovascular disease not listed under criterion 7), that would, in the opinion of the investigator, compromise the participant's safety or outcome in the trial; or lead to poor compliance with study visits and protocol requirements; or compromise the interpretation of trial safety and efficacy endpoints
16. Women who are currently pregnant or breast-feeding
17. Women of childbearing potential unwilling or unable to use appropriate effective contraception during the study intervention period and for at least 14 days after the last dose of study intervention; and unwilling to commit to refrain from donating eggs (ova, oocytes) for the purpose of reproduction during this period; definitions of childbearing potential and appropriate effective contraception given below**
18. Men who are unwilling to use a condom during the study period and for at least 90 days after the last dose of study drug during any activity that allows for the passage of ejaculate to another person; and are unwilling to commit to refrain from donating fresh unwashed semen
19. Known allergy to one or more of the study drugs
20. Taking a concomitant medication that has a known or predicted interaction with any of the study drugs to which the participant might be randomised. The participant need not be excluded if:

    1. the concomitant medication can be stopped or replaced with an alternative non-interacting medication, if needed AND
    2. the investigator judges there to be no residual clinical risk to the participant after stopping the concomitant medication (taking into account the washout period of 5x the half-life of the concomitant medication and the duration of the effect of the interaction on levels of study medication)
21. Taking a concomitant medication that is known to prolong the QTc interval. The participant need not be excluded if the concomitant medication can be stopped or replaced with an alternative medication, if needed, and the duration of the QTc prolongation is expected to resolve prior to dosing of study medication (taking into account the washout period of 5x the half-life of the concomitant medication)
22. Treatment with any immunosuppressive drugs within the 2 weeks prior to screening (taking systemic corticosteroids for less than 5 consecutive days and stopped at or prior to screening are not an exclusion; topical or inhaled steroids that are taken at a dose below the threshold considered to have systemic immunosuppressive effects are not excluded)
23. Participation in other clinical intervention trial with an investigational agent within 8 weeks prior to the first dosing day in this trial
24. 12-lead ECGs at screening or at baseline shows QTcF >450ms (men) or >460ms (women) calculated by Fridericia's formula; and/or any other clinically significant abnormality such as arrhythmia or ischaemia
25. Any of the following laboratory parameters at screening:

    1. Haemoglobin < 9g/dl
    2. Platelet count < 50 x 109 cells/L
    3. Absolute neutrophil count <1000 cells/μL
    4. Creatinine clearance of <75ml/min, calculated using Cockcroft-Gault equation*
    5. ALT or AST > 3 times the upper limit of normal
    6. Total bilirubin > 1.5 times upper limit of normal
    7. Serum potassium <3.5 mmol/L (not excluded if corrected to above this level)
    8. Serum magnesium < 0.70mmol/L (not excluded if corrected to above this level)
    9. Serum calcium (corrected for albumin level) < 2.10 mmol/L (not excluded if corrected to above this level)
26. Hepatitis B surface antigen positive (known, or on a test performed at screening)
27. HIV antibody positive (known, or on test performed at screening)*
28. Known Hepatitis C virus infection (unless also known to have negative PCR test)*

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-02-24 (Estimated); Study Completion 2027-08-11 (Estimated)

PRIMARY OUTCOMES:
Rate of change in log10(Time to Positivity of MGIT culture) (Phase 2B) | Over 0-12 weeks
  Primary Efficacy Outcome in Phase 2B, rate of change in log10(Time to positivity)
Favourable/Unfavourable outcome (Phase 2C) | at 48 weeks from randomisation
  Primary Efficacy Outcome in Phase 2C, the proportion of participants with a favourable outcome status

SECONDARY OUTCOMES:
Grade 3/4/5 adverse events (Phase 2B) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2B, grade 3/4/5 adverse events
Grade 3/4/5 adverse events (Phase 2C) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2C, grade 3/4/5 adverse events
Serious adverse events (Phase 2B) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2B, serious adverse events
Serious adverse events (Phase 2C) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2C, serious adverse events
Adverse events of special interest (Phase 2B) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2B, adverse events of special interest
Adverse events of special interest (Phase 2C) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2C, adverse events of special interest
Regimen-related adverse events (Phase 2B) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2B, Regimen-related adverse events
Regimen-related adverse events (Phase 2C) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2C, Regimen-related adverse events
Adverse events leading to withdrawal from the study (Phase 2B) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2B, Adverse events leading to withdrawal from the study
Adverse events leading to withdrawal from the study (Phase 2C) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2C, Adverse events leading to withdrawal from the study
Adverse events leading to discontinuation of the regimen (AESI) (Phase 2B) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2B, Adverse events leading to discontinuation of the regimen
Adverse events leading to discontinuation of the regimen (Phase 2C) | Up to 26 weeks from randomisation
  Safety outcome in Phase 2C, Adverse events leading to discontinuation of the regimen
Favourable/unfavourable status (Phase 2B) | At week 48
  Secondary Efficacy Outcome in Phase 2B, the proportion of participants with a favourable outcome status
Favourable/unfavourable status (Phase 2B) | At week 72
  Secondary Efficacy Outcome in Phase 2B and 2C, the proportion of participants with a favourable outcome status
Favourable/unfavourable status (Phase 2C) | At week 72
  Secondary Efficacy Outcome in Phase 2B and 2C, the proportion of participants with a favourable outcome status
Time to culture negative status (Phase 2B) | 0-24 weeks
  Secondary Efficacy Outcome in Phase 2B, time to culture negative status
Time to culture negative status (Phase 2C) | 0-24 weeks
  Secondary Efficacy Outcome in Phase 2C, time to culture negative status
Culture conversion measured from Mycobacterial Growth Indicator Tube system (MGIT) liquid culture results (Phase 2B) | weeks 4, 8, 12 and 16
  Secondary Efficacy Outcome in Phase 2B, culture conversion status
Culture conversion measured from Mycobacterial Growth Indicator Tube system (MGIT) liquid culture results (Phase 2C) | weeks 4, 8, 12 and 16
  Secondary Efficacy Outcome in Phase 2C, culture conversion status
PK parameters; Area under the plasma concentration versus time curve (AUC) over 0 to 24 hours | weeks 4 and 8
  Pharmacokinetic (PK) Outcomes; Area under the plasma concentration versus time curve (AUC) over 0 to 24 hours
PK parameters; Peak Plasma Concentration (CMax) | weeks 4 and 8
  Pharmacokinetic (PK) Outcomes; Peak Plasma Concentration (CMax)

CONTACTS AND LOCATIONS:
Locations (11):
- PMSI Institute of Pneumology "Chiril Draganiuc", Chisinau, Moldova
- South Africa (3):
  - TASK Brooklyn, Cape Town
  - University of Cape Town Lung Institute, Cape Town
  - TASK Eden, George
- Tanzania (3):
  - NIMR Mbeya, Mbeya
  - Kibong'oto Infectious Diseases Hospital, Moshi
  - NIMR Mwanza, Mwanza
- Uganda (2):
  - Joint Clinical Research Centre, Kampala
  - Makerere University Lung Institute, Kampala
- Vietnam (2):
  - National Lung Hospital, Hanoi
  - Pnth/Oucru, Ho Chi Minh City

REFERENCES:
- [Background] Eckhardt E, Li Y, Mamerow S, Schinkothe J, Sehl-Ewert J, Dreisbach J, Corleis B, Dorhoi A, Teifke J, Menge C, Kloss F, Bastian M. Pharmacokinetics and Efficacy of the Benzothiazinone BTZ-043 against Tuberculous Mycobacteria inside Granulomas in the Guinea Pig Model. Antimicrob Agents Chemother. 2023 Apr 18;67(4):e0143822. doi: 10.1128/aac.01438-22. Epub 2023 Mar 28. PMID 36975792
- [Background] Tenero D, Derimanov G, Carlton A, Tonkyn J, Davies M, Cozens S, Gresham S, Gaudion A, Puri A, Muliaditan M, Rullas-Trincado J, Mendoza-Losana A, Skingsley A, Barros-Aguirre D. First-Time-in-Human Study and Prediction of Early Bactericidal Activity for GSK3036656, a Potent Leucyl-tRNA Synthetase Inhibitor for Tuberculosis Treatment. Antimicrob Agents Chemother. 2019 Jul 25;63(8):e00240-19. doi: 10.1128/AAC.00240-19. Print 2019 Aug. PMID 31182528
- [Background] Li X, Hernandez V, Rock FL, Choi W, Mak YSL, Mohan M, Mao W, Zhou Y, Easom EE, Plattner JJ, Zou W, Perez-Herran E, Giordano I, Mendoza-Losana A, Alemparte C, Rullas J, Angulo-Barturen I, Crouch S, Ortega F, Barros D, Alley MRK. Discovery of a Potent and Specific M. tuberculosis Leucyl-tRNA Synthetase Inhibitor: (S)-3-(Aminomethyl)-4-chloro-7-(2-hydroxyethoxy)benzo[c][1,2]oxaborol-1(3H)-ol (GSK656). J Med Chem. 2017 Oct 12;60(19):8011-8026. doi: 10.1021/acs.jmedchem.7b00631. Epub 2017 Sep 27. PMID 28953378